CLINICAL TRIAL: NCT01068301
Title: A Phase I Pediatric Study of a Plerixafor Containing Regimen In Second Allogeneic Stem Cell Transplantation
Brief Title: A Pediatric Study of a Plerixafor Containing Regimen In Second Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOZBMT
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Chronic Myeloid Leukemia; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma
Keywords: Allogeneic Stem Cell transplantation; Plerixafor; Acute Lymphoblastic leukemia; Acute Myeloid leukemia; Chronic Myeloid leukemia; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma; Other Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Second Allogeneic Transplant Procedure Recipient (Other): Participants with Acute Lymphoblastic Leukemia (ALL); Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS); Chronic Myeloid Leukemia (CML); Juvenile Myelomonocytic Leukemia (JMML); Non-Hodgkin lymphoma (NHL) with evidence of bone marrow disease, receiving a second allogeneic transplant procedure.
  Intervention: Plerixafor
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — Plerixafor in combination with fludarabine, thiotepa and melphalan as a conditioning regimen for patients undergoing a second allogeneic transplant procedure (bone marrow or peripheral blood). A traditional 3+3 phase I design will be employed during this study, where dose escalations are planned in groups of 3 participants. No intra-participant escalation will be allowed and dose escalation will not be considered until toxicity information is available from at least 3 evaluable participants at the current dose level.Plerixafor will be given intravenously (IV) rather than subcutaneously (SQ) to minimize discomfort associated with repeated daily injections (up to 3) to the pediatric population of this study.
  Other Names: AMD3100; Mozobil®

SUMMARY:
Patients with refractory hematologic malignancies, including those who develop recurrent disease after allogeneic hematopoietic stem cell transplantation (HSCT) have a dismal prognosis. Historically, both regimen-related mortality and disease recurrence have been significant causes of treatment failure in this heavily pre-treated patient population. Novel therapeutic agents that target molecular signaling mechanisms and increase the sensitivity of leukemic cells to apoptosis may clearly play a role in this setting.

This study hypothesizes that interrupting the SDF-1/CXCR4 axis using the selective CXCR4 antagonist plerixafor may be useful as a leukemic stem cell mobilizing agent for patients who are refractory to standard dose chemotherapy and in relapse after an allogeneic transplant. This hypothesis is based on the dependence of leukemia cells on MSCs for survival signals as described above and on the preclinical data that suggest increased efficacy by antileukemia agents when leukemia cells are separated from MSCs.

In the present trial, the study proposes to add plerixafor to enhance the conditioning regimen cytotoxicity. At this time the goal is to determine the maximum tolerated dose (MTD) of plerixafor through the process of dose limiting toxicity (DLT) evaluation. Pharmacokinetic studies will be conducted. Additional studies will quantify and the content of leukemia cells and key regulatory and effector T cell populations in the bone marrow and blood before and after exposure to this medication.

If the observed outcomes of this trial are promising, it could serve as a platform on which to study further use of plerixafor as a complimentary agent with conditioning as well as other chemotherapeutic regimens for patients with relapsed or refractory hematologic malignancies.

DETAILED DESCRIPTION:
This study will determine the following objectives:

1. To determine the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of plerixafor in combination with fludarabine, thiotepa, and melphalan as a conditioning regimen for children and young adults undergoing a second allogeneic stem cell transplant (SCT) procedure.
2. The study determines the secondary objectives:

   * To describe the pharmacokinetic properties of plerixafor in this study population
   * To estimate the cumulative incidence of relapse and overall survival in study participants at one year after this second transplant procedure
3. Other exploratory objectives include:

   * To study the correlation between the pharmacokinetic properties of plerixafor and key regulatory and effector T cell populations in blood before and after exposure to plerixafor.
   * To evaluate the content of leukemia cells in bone marrow and in blood before and after exposure to plerixafor
   * To evaluate key regulatory and effector T cell populations in bone marrow and in blood before and after exposure to plerixafor

ELIGIBILITY:
Inclusion Criteria:

* Age less than or equal to 21 years old.
* One of the following hematologic malignancies that has relapsed after prior allogeneic hematopoietic stem cell transplantation:
* Acute lymphoblastic leukemia (ALL)
* Acute myeloid leukemia (AML)
* Myelodysplastic syndrome (MDS)
* Chronic myeloid leukemia (CML)
* Juvenile myelomonocytic leukemia (JMML)
* Non-Hodgkin's lymphoma (NHL) with evidence of bone marrow disease
* Has a suitable human leukocyte antigen (HLA) matched family member or unrelated donor available for stem cell donation. A "matched" donor is defined as matching at 5/6 or 6/6 HLA loci.
* Does not have active central nervous system (CNS) malignancy (history of CNS disease allowed).
* No prior neuromuscular dysfunction or all prior grade I-IV neuromuscular dysfunctions have subsided > 4 weeks prior to enrollment.
* Cardiac shortening fraction greater than or equal to 25%.
* Creatinine clearance greater than or equal to 50 ml/min/1.73 m2
* Forced vital capacity (FVC) greater than or equal to 40% of predicted value or pulse oximetry greater than or equal to 92% on room air.
* Karnofsky or Lansky (age-dependent) performance score of greater than or equal to 50 .
* Off all treatment for acute or chronic graft-versus-host disease (GVHD) for at least 7 days prior to the initiation of conditioning.
* Bilirubin less than or equal to 3 times the upper limit of normal for age.
* Alanine aminotransferase (ALT) less than or equal to 3.0 times the upper limit of normal for age.
* White blood cell count of less than 50,000/mm3
* Not pregnant as confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment.
* Not lactating.
* All patients of childbearing potential must agree to use an effective birth control method

Exclusion Criteria:

* Pregnant and lactating females are excluded from participation as the short and long-term effects of the preparative agents and infusion on a fetus and a nursing child through breast milk are not entirely known at this time.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2010-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To determine the dose-limiting toxicity and maximum tolerated dose of plerixafor in combination with fludarabine, thiotepa and melphalan as a conditioning regimen for patients undergoing a second allogeneic transplant procedure. | 7 days post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Srinivasan, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org